CLINICAL TRIAL: NCT03877861
Title: Validation of Readiband™ Actigraph and Associated Sleep/Wake Classification Algorithms in Predicting Cancer Related Fatigue and Diseases Progression in High Grade Glioma
Brief Title: Validation of Readiband™ Actigraph and Associated Sleep/Wake Classification Algorithms
Status: Completed | Type: Observational
Sponsor: Allina Health System (Other)
Responsible Party: Sponsor
Other Study IDs: NSJT-1701
Record Dates: First submitted 2018-03-14; First posted 2019-03-18 (Actual); Last update posted 2021-06-09 (Actual); Status verified 2021-06

CONDITIONS: Glioma; Glioblastoma
MeSH Terms: conditions — Glioma; Glioblastoma

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: Yes | US Export: No

GROUPS / COHORTS (2):
- Readiband Sleep Tracking - Patient: This group is comprised of 25 participants with a diagnosis of primary Grade IV glioma. A Readiband™ Sleep Tracker device will be provided to each participant, along with necessary instructions. Participantswill return home with the device and fatigue data will be obtained from the device at subsequent standard care follow-up visits.
  Interventions: Device: Readiband Sleep Tracking
- Readiband Sleep Tracking - Control: Aggregate fatigue data and sleep patterns for a group of 30 healthy controls procured from FatigueScience in a de-identified manner for data analysis purposes.
  Interventions: Device: Readiband Sleep Tracking

INTERVENTIONS:
Device: Readiband Sleep Tracking — Once a patient has consented to study progression, a Readiband™ Sleep Tracker device will be provided to the patient, along with necessary instructions. Patients will return home with the device and fatigue data will be obtained from the device at subsequent standard care follow-up visits. In addition, surveys related to fatigue and quality of life will be administered via secure electronic survey to participants.

SUMMARY:
This pilot study will assess feasibility and to obtain initial estimates of efficacy of Sleep Activity and Task Effectiveness (SAFTE) model, which can accurately estimate the impact of scheduling factors and sleep history on both safety and productivity. The SAFTE model will be used to asses cancer-related fatigue and study potential associations of change in sleep patterns to tumor recurrence in patients with high grade glioma. Data will be collected using the Readiband™ Sleep Tracker (https://www.fatiguescience.com/sleep-science-technology/). The Readiband device captures high-resolution sleep data, validated against the clinical gold standard of polysomnography with 92% accuracy. Sleep data is transmitted to the cloud automatically for SAFTE Fatigue Model analysis. We will correlate clinical progression data obtained from the patient's electronic medical record with SAFTE data.

ELIGIBILITY:
Inclusion Criteria

i. Patients aged between 22 and 70. ii. Patients must have a histologic diagnosis of primary Grade IV glioma. iii. Patients must have received maximal debulking surgery and radiotherapy concomitant with Temozolomide (≥ 75% of their recommended temozolomide dosage is required).

iv. Patients with KPS ≥70. v. Life expectancy at least 3 months. vi. Patients must have signed informed consent for study participation. vii. Patients should be English speakers.

Exclusion Criteria

i. Patients enrolled in active clinical treatment trials for primary Grade IV glioma.

ii. Patients with progressive disease after completion of radiotherapy concomitant with Temozolomide as per RANO criteria. Suspected pseudoprogression should be confirmed by additional imaging studies ordered as part of standard care.

iii. Patients with known other active malignancy diagnosed in the past 3 years (except for in situ malignancies).

iv. Patients who are pregnant or trying to get pregnant. v. Patients unable to wear the ReadiBand device continuously during study duration.

vi. Patients with infra-tentorial tumors. vii. Patients with known psychiatric concerns. viii. Significant co-morbidities at baseline which would prevent maintenance Temozolomide treatment:

1. Thrombocytopenia (platelet count < 100 x 103/μL)
2. Neutropenia (absolute neutrophil count < 1.5 x 103/μL)
3. CTC grade 4 non-hematological Toxicity (except for alopecia, nausea, vomiting)
4. Significant liver function impairment - AST or ALT > 3 times the upper limit of normal
5. Total bilirubin > upper limit of normal, if clinically significant
6. Significant renal impairment (serum creatinine > 1.7 mg/dL)

Ages: 22 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients with Grade IV gliomas treated at Abbott Northwestern Hospital's Givens Brain Tumor Center will comprise the study population. Patients enrolled in this study must intend to complete post-surgery chemoradiation as part of their standard treatment. Twenty-five patients will prospectively be included in the study. Aggregate fatigue data and sleep patterns for a group of 30 healthy controls will be procured from FatigueScience in a de-identified manner for data analysis purposes.
Sampling Method: Non-Probability Sample
Enrollment: 7 (Actual)
Dates: Start 2018-03-15 (Actual); Primary Completion 2021-05-01 (Actual); Study Completion 2021-05-01 (Actual)

PRIMARY OUTCOMES:
Correlation between sleep patterns and disease progression/recurrence | Participant enrollment to 12 months (or until tumor progression)
  An estimate of correlation between sleep patterns in the brain tumor patient population and disease progression or recurrence compared to those of the general population.

SECONDARY OUTCOMES:
Correlation between SAFTE fatigue predictions and self-reported fatigue levels | Participant enrollment to 12 months (or until tumor progression)
  An estimate of correlation between SAFTE fatigue predictions and self-reported fatigue levels in patients with GBM
Sleep pattern differences between healthy controls and brain tumor patients | Participant enrollment to 12 months (or until tumor progression)
  Comparison of differences in sleep patterns in brain tumor patients to those of the general population.
Correlation between fatigue and sleep patterns and treatment tolerance/success | Participant enrollment to 12 months (or until tumor progression)
  An estimate of correlation between fatigue and sleep patterns and treatment tolerance/success, as determined by MRI imaging and RANO criteria.
Change in Sleep, Activity, Fatigue, and Task Effectiveness (SAFTE) score | Participant enrollment to 12 months (or until tumor progression)

CONTACTS AND LOCATIONS:
Overall Officials: John Trusheim, MD, Principal Investigator — Allina Health
Locations (1):
- Abbott Northwestern Hospital, Minneapolis, Minnesota, United States

IPD SHARING:
Plan to Share IPD: No